CLINICAL TRIAL: NCT01565616
Title: A Phase II Study of Hematopoietic Stem Cell Therapy for Young Adults With Severe Sickle Cell Disease
Brief Title: Bone Marrow Transplantation in Young Adults With Severe Sickle Cell Disease
Acronym: STRIDE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Lakshmanan Krishnamurti, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00068287; 1R34HL108761-01 (NIH)
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-10

CONDITIONS: Sickle Cell Disease
Keywords: Severe Sickle Cell Disease; Hematopoietic cell transplantation (HCT); Hematopoietic Stem Cell Therapy; Bone Marrow Transplant; Hematologic Diseases; Genetic Diseases; Anemia; Hemolytic; Congenital; Human Leukocyte Antigen; HLA
MeSH Terms: conditions — Anemia, Sickle Cell; Hematologic Diseases; Genetic Diseases, Inborn; Anemia; Hemolysis | interventions — Transplantation Conditioning; Bone Marrow Transplantation; Busulfan; fludarabine; fludarabine phosphate; Antilymphocyte Serum; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bone Marrow Transplant Recipients (Experimental): Adults with sickle cell disease undergoing a bone marrow transplant from an HLA-identical sibling donor or an unrelated HLA-matched donor.
  Interventions: Drug: Conditioning Regimen with Bone Marrow Transplant

INTERVENTIONS:
Drug: Conditioning Regimen with Bone Marrow Transplant — The bone marrow transplant regimen is below. Day 0 is the day of the transplant. The - sign is the number of days before and the + sign is the number of days after the transplant.
  Day -8 BU 3.2 mg/ kg/dose IV
  Day -7 BU 3.2 mg/kg/dose IV, FLU 35mg/m2 IV
  Day -6 BU 3.2 mg/kg/dose IV, FLU 35mg/m2 IV, ATG 0.5mg/kg IV
  Day -5 BU 3.2 mg/kg/dose IV, FLU 35mg/m2 IV, ATG 1.0mg/kg IV
  Day -4 FLU 35mg/m2 IV, ATG 1.5mg/kg IV
  Day -3 FLU 35mg/m2 IV, ATG 1.5mg/kg IV
  Day -2 ATG 1.5mg/kg IV
  Day -1 Rest
  Day 0 Stem cell infusion
  Graft Versus Host Disease (GVHD) Regimen
  Day -3 Calcineurin Inhibitor (Cyclosporine or Tacrolimus) therapeutic doses through day 180, then taper
  Day 0 Stem cell infusion
  Day +1 Methotrexate 7.5 mg/m2 IV
  Day +3 Methotrexate 7.5 mg/m2 IV
  Day +6 Methotrexate 7.5 mg/m2 IV
  Day+11 Methotrexate 7.5 mg/m2 IV
  Other Names: Busulfan (BU); Myleran; Busulfex IV; Fludarabine (FLU); Fludara; Rabbit Anti-thymocyte globulin (ATG); Thymoglobulin

SUMMARY:
This is a Phase II, single arm, multi-center trial. It is designed to estimate the efficacy and toxicity of hematopoietic stem cell transplantation (HSCT) in patients with sickle cell disease (SCD) who have high risk features.

The primary goal of this multi-center Phase II study is to determine the safety and feasibility of a conditioning regimen consisting of busulfan (Bu)/ fludarabine (Flu)/ anti-thymocyte globulin (ATG) in adult patients with severe SCD. A two-component design will be used for this study. The first component will be restricted to patients who have an HLA-identical sibling donor. Five patients will be transplanted during the first component of the study. If no more than 2 of the first 5 patients experience unacceptable toxicity, including death, within the first six months after transplantation, then the safety of the regimen will be considered promising in adult SCD patients.

The second component will include patients who have a related or an unrelated human leukocyte antigen (HLA) matched donor. Up to 15 additional patients will be transplanted in this component of the study which will evaluate the safety and feasibility of unrelated donor hematopoietic cell transplantation (HCT) in adults with SCD. Data related to study endpoints for 1 year after transplantation will be collected; however, participating centers will be encouraged to conduct long-term follow-up evaluations of patients according to standard institutional guidelines. The purpose of this pilot safety trial is to see if this approach is feasible and meets accrual goals lending support to the development of a subsequent full scale investigation of HCT and comparing outcomes in a transplantation cohort to a control cohort of adults eligible for, but unwilling or unable to receive HCT treated by supportive therapy with a primary endpoint of five years survival for this full scale comparative trial.

DETAILED DESCRIPTION:
This is a Phase II, single arm, multi-center trial. It is designed to estimate the efficacy and toxicity of hematopoietic stem cell transplantation (HSCT) in patients with sickle cell disease (SCD) who have high risk features.

The primary goal of this multi-center Phase II study is to determine the safety and feasibility of a conditioning regimen consisting of busulfan (Bu)/ fludarabine (Flu)/ anti-thymocyte globulin (ATG) in adult patients with severe SCD. A two-component design will be used for this study. The first component will be restricted to patients who have an HLA-identical sibling donor. Five patients will be transplanted during the first component of the study. If no more than 2 of the first 5 patients experience unacceptable toxicity, including death, within the first six months after transplantation, then the safety of the regimen will be considered promising in adult SCD patients.

The second component will include patients who have a related or an unrelated human leukocyte antigen (HLA) matched donor. Up to 15 additional patients will be transplanted in this component of the study which will evaluate the safety and feasibility of unrelated donor hematopoietic cell transplantation (HCT) in adults with SCD. Data related to study endpoints for 1 year after transplantation will be collected; however, participating centers will be encouraged to conduct long-term follow-up evaluations of patients according to standard institutional guidelines. The purpose of this pilot safety trial is to see if this approach is feasible and meets accrual goals lending support to the development of a subsequent full scale investigation of HCT and comparing outcomes in a transplantation cohort to a control cohort of adults eligible for, but unwilling or unable to receive HCT treated by supportive therapy with a primary endpoint of five years survival for this full scale comparative trial.

The primary objective is to determine event-free survival (EFS) at 1 year after hematopoietic cell transplantation (HCT) using bone marrow in patients with sickle cell disease. Death, disease recurrence or graft rejection by 1 year will be considered events for this endpoint.

Secondary objectives include determining the effect of HCT on clinical and laboratory manifestations of severe sickle cell disease and determining the incidence of other transplant-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe sickle cell disease and have one or more of the following:

  1. Clinically significant neurologic event (stroke) or any neurological deficit lasting > 24 hours
  2. History of two or more episodes of acute chest syndrome (ACS) in the 2-year period preceding enrollment despite the institution of supportive care measures (i.e. asthma therapy and/or hydroxyurea). Acute Chest Syndrome (ACS) is defined as new pulmonary alveolar consolidation (or infiltrate) involving at least one complete lung segment associated with acute symptoms including one or more of the following: fever ≥ 38.5 Celsius, chest pain, tachypnea per age adjusted normal, intercostal retractions/nasal flaring/use of accessory muscles of respiration, wheezing, rales or cough that is not attributed to asthma or bronchiolitis.
  3. History of three or more severe pain crises per year in the 2-year period preceding enrollment despite the institution of supportive care measures (i.e. a pain management plan and/or treatment with hydroxyurea). Pain Crisis is defined as new onset of pain that last for at least 2 hours for which there is no other explanation (i.e. vaso-occlusive, priapism).
  4. Administration of regular red blood cell (RBC) transfusion therapy, defined as receiving 8 or more transfusions per year for greater than or equal to 1 year to prevent vaso-occlusive clinical complications (i.e. pain, stroke, and acute chest syndrome)
  5. Trans-thoracic echocardiograph evidence of tricuspid valve regurgitant jet (TRJ) velocity greater than or equal to 2.7 m/sec.
* Adequate physical function as measured by:

  1. Karnofsky performance score greater than or equal to 60
  2. Cardiac function: Left ventricular ejection fraction (LVEF) > 40%; or LV shortening fraction > 26% by cardiac echocardiogram or by multigated acquisition (MUGA) scan.
  3. Pulmonary function: Pulse oximetry with a baseline O2 saturation of greater than or equal to 85% and diffusing capacity of the lungs for carbon monoxide (DLCO) > 40% (corrected for hemoglobin)
  4. Renal function: Serum creatinine ≤ 1.5 x upper limit of normal for age and 24-hour urine creatinine clearance > 70 mL/min/1.73 m2 by radionuclide glomerular filtration rate (GFR); or GFR > 70 mL/min/1.73 m2 by radionuclide GFR.
  5. Hepatic function: Serum conjugated (direct) bilirubin < 2x upper limit of normal for age as per local laboratory; and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 5 times upper limit of normal as per local laboratory. Patients whose hyperbilirubinemia is the result of hyperhemolysis, or a severe drop in hemoglobin post blood transfusion, are not excluded
  6. If the patient has been receiving chronic transfusion therapy for greater than or equal to 1 year and has clinical evidence of iron overload by serum ferritin (mean of 3 ferritin levels >1000 and chronic transfusions >20 in a lifetime or MRI), evaluation by liver biopsy is required. Histological examination of the liver must document the absence of cirrhosis, bridging fibrosis and active hepatitis. The absence of bridging fibrosis will be determined using the histological grading and staging scale as described by Ishak and colleagues (1995).
* Patients must have a related or unrelated bone marrow donor with HLA-matched at 8 of 8 HLA-A, B, C, and DRB1 loci by allelic testing. Umbilical cord blood or peripheral blood stem cell donors will not be accepted.

Exclusion Criteria:

* Patients with cirrhosis of the liver, uncontrolled bacterial, viral or fungal infection in the 6 weeks before enrollment, or seropositivity for HIV
* Patients who have received prior HCT
* Patients who within 3 months of enrollment have participated in another clinical trial in which the patient received an investigational drug or device or off-label use of a drug or device
* Patients who demonstrate lack of compliance with prior medical care
* Patients who are unwilling to use approved contraception for at least 6 months after transplant
* Patients who have a history of substance abuse in the last 5 years that interferes with their care
* Patients who are pregnant or breast feeding
* Patients unable to provide consent

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmanan Krishnamurti, MD, Principal Investigator — Emory University
Locations (8):
- United States (8):
  - Children's Hospital of Oakland, Oakland, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Duke University Medical Center, Durham, North Carolina
  - Chidren's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 8 study locations between March, 2012 and June, 2015.
Pre-assignment Details: The first component of the study was restricted to 5 patients with a related donor. If no more than 2 of the first 5 patients experienced unacceptable toxicity within six months of transplantation then the safety of the regimen was considered promising and the study could include patients with a related or unrelated HLA matched donor.
Groups:
- Bone Marrow Transplant Recipients: Individuals with severe sickle cell disease receiving hematopoietic cell transplantation (HCT) from a human leukocyte antigen (HLA)-identical sibling donor or an unrelated HLA-matched donor
Period: Overall Study
Arm/Group | Bone Marrow Transplant Recipients
Started | 22
First Component: 5 Related Donors (The first component was restricted to patients having an HLA-identical sibling donor.) | 5
Second Component: Related or Unrelated (The second component included patients having a related or unrelated HLA matched donor.) | 17
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Individuals with severe sickle cell disease receiving hematopoietic cell transplantation (HCT) from a human leukocyte antigen (HLA)-identical sibling donor or an unrelated HLA-matched donor
Groups:
- Bone Marrow Transplant Recipients: Individuals receiving a bone marrow transplant at one of 10 study locations, between March 2012 and June, 2015.
Arm/Group | Bone Marrow Transplant Recipients
Number analyzed (Participants) | 22
Age, Customized [Count of Participants; unit: Participants]
  16-19 years of age | 6
  20-24 years of age | 8
  24-29 years of age | 6
  30-40 years of age | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22
Donor Relation [Count of Participants; unit: Participants]
  Related | 17
  Unrelated | 5
Indication of Severe Sickle Cell Disease [Count of Participants; unit: Participants] — Participants were eligible for the study if they had one or more of the following:
  * Significant neurological event, such as a stroke or any neurological deficit lasting longer than 24 hours
  * History of acute chest syndrome (ACS)
  * History of 3 or more pain crises per year
  * Regular red blood cell (RBC) transfusions (8 or more per year)
  * Trans-thoracic echocardiographic evidence of tricuspid valve regurgitant jet (TRJ) velocity 2.7 m/sec
  Participants
    Significant neurological event (stroke) | 2
    Acute chest syndrome | 2
    Recurrent pain events | 15
    Regular RBC transfusion therapy | 4
    Elevated TRJ Velocity | 4

OUTCOME MEASURES:

1. Primary Outcome: Event -Free Survival Rate
Description: Event-free survival is defined as stable donor erythropoiesis with no new clinical evidence of sickle cell disease. Primary or late graft rejection, disease recurrence, and death are considered events for this endpoint.
Time Frame: 1 year after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant Recipients
Number analyzed (Participants) | 22
Participants | 19

2. Secondary Outcome: Graft Failure
Description: Primary graft failure occurs when a transplant recipient does not achieve donor chimerism following a bone marrow transplant. Secondary graft failure occurs when graft fails after donor chimerism had initially occurred.
Time Frame: 1 year after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant Recipients
Number analyzed (Participants) | 22
Participants
  Primary graft failure | 0
  Secondary graft failure | 1

3. Secondary Outcome: Acute Graft Versus Host Disease (GVHD)
Description: Acute GVHD was graded according to the Center for International Blood and Marrow Transplant Research (CIBMTR) consensus criteria. Clinical manifestations of acute GVHD include skin, liver, and gastrointestinal symptoms. Grading of acute GVHD is determined by size of maculopapular rash, bilirubin and stool output. Acute GVHD grades range from 0 to 4 with 0 indicating no GVHD and 4 representing the most severe grade.
  Grade II is defined as a maculopapular rash over 25-50% of body surface area (BSA), bilirubin of 3.1 to 6 mg/dL, and stool output of 1000-1500 mL/d (for adults).
  Grade III is defined as a maculopapular rash over more than 50% of BSA, bilirubin of 6.1 to 15 mg/dL, and stool output of greater than 1500 mL/d (for adults).
  Grade IV is defined as generalized erythroderma with bullous formation, bilirubin greater than 15 mg/dL, and severe abdominal pain with or without ileus.
Time Frame: 1 year after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant Recipients
Number analyzed (Participants) | 22
Participants
  Grade II Acute GVHD | 3
  Grade III Acute GVHD | 1
  Grade IV Acute GVHD | 0

4. Secondary Outcome: Chronic Graft Versus Host Disease (GVHD)
Description: Chronic GVHD was graded according to the National Institutes of Health (NIH) 2014 Consensus Criteria Diagnosis and scoring the severity of chronic GVHD is determined by evaluating symptoms of the skin, nails, hair, mouth, eyes, genitalia, gastrointestinal tract, liver, lungs, muscles, fascia and joints, immune function as well as other symptoms such as ascites and neuropathy. Chronic GVHD is graded as mild, moderate or severe based on the number of organ sites impacted and the severity of symptoms.
Time Frame: 1 year after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant Recipients
Number analyzed (Participants) | 22
Participants
  Mild Chronic GVHD | 3
  Moderate Chronic GVHD | 2
  Severe Chronic GVHD | 1

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as survival with or without sickle cell disease after hematopoietic cell transplantation (HCT).
Time Frame: 1 year after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant Recipients
Number analyzed (Participants) | 22
Participants | 20

6. Secondary Outcome: Time to Neutrophil and Platelet Engraftment
Description: Time to neutrophil engraftment is defined as the first of 3 measurements on different days when the patient has an absolute neutrophil count of at least 500/µL after conditioning. Time to Platelet engraftment is defined as the first day of a minimum of 3 measurements on different days that the patient has achieved a platelet count > 50,000/µL, without receiving a platelet transfusion in the previous 7 days.
Time Frame: 1 year after transplant
Measure: Median (Full Range); unit: Days
Arm/Group | Bone Marrow Transplant Recipients
Number analyzed (Participants) | 22
Days
  Neutrophil engraftment | 17 [12 to 26]
  Platelet | 21 [13 to 26]

7. Secondary Outcome: Transplant Related Outcomes
Description: Common transplant related complications were monitored as a secondary outcome measure of this study. These transplant related complications include hepatic veno-occlusive disease (VOD), idiopathic pneumonia syndrome (IPS), central nervous system (CNS) toxicity complications of posterior reversible encephalopathy syndrome (PRES), hemorrhage, and seizures, cytomegalovirus (CMV) infection, adenovirus infection, Epstein-Barr virus (EBV) infection, post-transplant lymphoproliferative disease (PTLD), and invasive fungal infection.
Time Frame: 1 year after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant Recipients
Number analyzed (Participants) | 22
Participants
  Hepatic Veno-occlusive Disease (VOD) | 0
  Idiopathic Pneumonia Syndrome (IPS) | 1
  PRES | 1
  Central Nervous System Toxicity: Hemorrhage | 1
  Central Nervous System Toxicity: Seizure | 1
  Cytomegalovirus (CMV) Infection | 11
  Adenovirus Infection | 0
  Epstein-Barr Virus (EBV) Infection | 4
  Post-transplant Lymphoproliferative Disease | 1
  Invasive Fungal Infection | 0

8. Post Hoc Outcome: PROMIS-57 Scores Health Related Quality of Life
Description: Health related quality of life was measured with the 57 item Patient-Reported Outcomes Measurement Information System (PROMIS-57). The PROMIS-57 includes 8 domains of health. The domains of Anxiety, Depression, Fatigue, Pain Interference, Physical Function, Satisfaction with Social Role, and Sleep Disturbances each include 8 items. Respondents indicate the degree to which statements about specific health issues are problematic on a scale of 1 to 5 and responses are converted to a t-score metric. A score of 50 is the mean score for the general population in the United States, with a standard deviation of 10. Scores above 50 indicate the topic of the domain is being experienced more than average while scores below 50 mean that it is less than average.
  The domain of Pain Intensity is measured with a single item asking participants to rate their average pain on a scale from 0 (no pain) to 10 (worst imaginable pain). The raw mean score is used.
Time Frame: Baseline, 1 year after transplant
Population: This outcome measure compared quality of life scores one year post-HCT to baseline in the 17 participants who completed the surveys.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bone Marrow Transplant Recipients
Number analyzed (Participants) | 17
units on a scale
  Anxiety domain score: baseline | 50.6 (10.4)
  Anxiety domain score: 1 year: number analyzed (Participants) | 16
  Anxiety domain score: 1 year | 48.1 (10.5)
  Depression domain score: baseline | 44.7 (6.7)
  Depresssion domain score: 1 year: number analyzed (Participants) | 16
  Depresssion domain score: 1 year | 46.9 (10.3)
  Fatigue domain score: baseline | 48.0 (10.5)
  Fatigue domain score: 1 year: number analyzed (Participants) | 16
  Fatigue domain score: 1 year | 46.1 (13.4)
  Pain interference domain score: baseline | 58.5 (10.3)
  Pain interference domain score: 1 year: number analyzed (Participants) | 16
  Pain interference domain score: 1 year | 50.1 (11.6)
  Physical function domain score: baseline | 44.1 (8.0)
  Physical function domain score: 1 year: number analyzed (Participants) | 16
  Physical function domain score: 1 year | 50.1 (11.0)
  Social role satisfaction domain score: baseline | 51.7 (11.6)
  Social role satisfaction domain score: 1 year: number analyzed (Participants) | 16
  Social role satisfaction domain score: 1 year | 52.4 (12.3)
  Sleep disturbance domain score: baseline | 47.7 (11.9)
  Sleep disturbance domain score: 1 year: number analyzed (Participants) | 16
  Sleep disturbance domain score: 1 year | 46.9 (9.6)
  Pain intensity domain score: baseline | 3.2 (3.4)
  Pain intensity domain score: 1 year: number analyzed (Participants) | 16
  Pain intensity domain score: 1 year | 2.4 (3.0)
Statistical Analysis 1: Comparison: Bone Marrow Transplant Recipients; This statistical analysis is the paired difference in t-scores of the anxiety domain of the PROMIS-57 quality of life scale. 16 participants with paired measurements of the PROMIS-57 survey (baseline and 1 year) are included in this analysis; Test type: Other; p = 0.52, t-test, 2 sided; Mean Difference (Net) = -1.7, Standard Deviation 10.4
Statistical Analysis 2: Comparison: Bone Marrow Transplant Recipients; This statistical analysis is the paired difference in t-scores of the depression domain of the PROMIS-57 quality of life scale. 16 participants with paired measurements of the PROMIS-57 survey (baseline and 1 year) are included in this analysis; Test type: Other; p = 0.12, t-test, 2 sided; Mean Difference (Net) = 2.7, Standard Deviation 6.4
Statistical Analysis 3: Comparison: Bone Marrow Transplant Recipients; This statistical analysis is the paired difference in t-scores of the fatigue domain of the PROMIS-57 quality of life scale. 16 participants with paired measurements of the PROMIS-57 survey (baseline and 1 year) are included in this analysis; Test type: Other; p = 0.54, t-test, 2 sided; Mean Difference (Net) = -1.3, Standard Deviation 8.5
Statistical Analysis 4: Comparison: Bone Marrow Transplant Recipients; This statistical analysis is the paired difference in t-scores of the pain interference domain of the PROMIS-57 quality of life scale. 16 participants with paired measurements of the PROMIS-57 survey (baseline and 1 year) are included in this analysis; Test type: Other; p = 0.006, t-test, 2 sided; Mean Difference (Net) = -7.5, Standard Deviation 9.3
Statistical Analysis 5: Comparison: Bone Marrow Transplant Recipients; This statistical analysis is the paired difference in t-scores of the physical function domain of the PROMIS-57 quality of life scale. 16 participants with paired measurements of the PROMIS-57 survey (baseline and 1 year) are included in this analysis; Test type: Other; p = 0.044, t-test, 2 sided; Mean Difference (Net) = 5.8, Standard Deviation 10.5
Statistical Analysis 6: Comparison: Bone Marrow Transplant Recipients; This statistical analysis is the paired difference in t-scores of the satisfaction with social role domain of the PROMIS-57 quality of life scale. 16 participants with paired measurements of the PROMIS-57 survey (baseline and 1 year) are included in this analysis; Test type: Other; p = 0.85, t-test, 2 sided; Mean Difference (Net) = 0.6, Standard Deviation 11.8
Statistical Analysis 7: Comparison: Bone Marrow Transplant Recipients; This statistical analysis is the paired difference in t-scores of the sleep disturbances domain of the PROMIS-57 quality of life scale. 16 participants with paired measurements of the PROMIS-57 survey (baseline and 1 year) are included in this analysis; Test type: Other; p = 0.88, t-test, 2 sided; Mean Difference (Net) = 0.5, Standard Deviation 13.5
Statistical Analysis 8: Comparison: Bone Marrow Transplant Recipients; This statistical analysis is the paired difference in raw scores of the pain intensity domain of the PROMIS-57 quality of life scale. 16 participants with paired measurements of the PROMIS-57 survey (baseline and 1 year) are included in this analysis; Test type: Other; p = 0.53, t-test, 2 sided; Mean Difference (Net) = -0.5, Standard Deviation 3.1

ADVERSE EVENTS:
Time Frame: Data on adverse events were collected from when the patient consented to participate in the study through 1 year after hematopoietic cell transplantation (HCT).
Arm/Group | Bone Marrow Transplant Recipients
All-Cause Mortality (participants affected / at risk) | 2/22
Serious Adverse Events (participants affected / at risk) | 14/22
Other Adverse Events (participants affected / at risk) | 12/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone Marrow Transplant Recipients (N=22)
Hospitalization due to abdominal pain, diarrhea, and bloody stools (Gastrointestinal disorders) | 1 (1)
Hospitalization due to abdominal pain, nausea, vomiting, and elevated liver enzymes (Gastrointestinal disorders) | 1 (1)
Hospitalization due to acute inflammatory bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalization due to acute on chronic pain (General disorders) | 1 (1)
Anemia secondary to hemolysis (Blood and lymphatic system disorders) | 1 (1)
Hospitalization due to chest pain, secondary to pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Elevated liver enzymes (Hepatobiliary disorders) | 2 (3)
Hospitalization due to elevated prograf level (Surgical and medical procedures) | 1 (1)
Hospitalization due to exacerbation of pain syndrome (General disorders) | 1 (1)
Facial swelling with sore throat (General disorders) | 1 (1)
Hospitalization due to fever, malaise, and chills (Infections and infestations) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1)
Gallstones with hyperbilirubinemia (Hepatobiliary disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (2)
Generalized pain (General disorders) | 1 (1)
Headache requiring Norco (General disorders) | 1 (1)
Hemolysis with rising creatinine (Blood and lymphatic system disorders) | 1 (1)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 2 (2)
Mucosistis, esophageal pain, and low back pain (General disorders) | 1 (1)
Neurological changes (Nervous system disorders) | 2 (2)
Opioid-induced over-sedation (Injury, poisoning and procedural complications) | 1 (1)
Hospitalization due to pain crisis (Blood and lymphatic system disorders) | 1 (1)
Hospitalization due to pericardial effusion (Cardiac disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1)
Hospitalization due to persistent fever (General disorders) | 1 (1)
Hospitalization due to pneumonia with hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PRES with intercerebral hemorrhage associated with severe hypertension (Vascular disorders) | 1 (1)
Prograf toxicity (Surgical and medical procedures) | 1 (1)
Hospitalization due to progressive respiratory distress with hypoxemia (Blood and lymphatic system disorders) | 1 (1)
Removal of central venous catheter due to possible thrombus (Blood and lymphatic system disorders) | 1 (1)
Respiratory distress secondary to large pharyngeal blood clot (Blood and lymphatic system disorders) | 1 (1)
Hospitalization due to seizure and infection (Infections and infestations) | 1 (1)
Hospitalization due to severe nausea, vomiting and diarrhea (Gastrointestinal disorders) | 1 (1)
Urinary retention, dysuria, and hesitancy (Renal and urinary disorders) | 1 (1)
Vascular disorder with facial swelling (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone Marrow Transplant Recipients (N=22)
Alopecia (Immune system disorders) | 1 (1)
Anorexia (General disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchiolitis obliterans (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Cranial Bell's Palsy (Nervous system disorders) | 1 (1)
Deep bone pain (General disorders) | 1 (1)
Diabetes mellitus (Endocrine disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Elevated alkaline phosphatase (Hepatobiliary disorders) | 1 (1)
Elevated alanine transaminase (Hepatobiliary disorders) | 2 (2)
Extremity pain (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Reduced hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Central nervous system hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Hyperglycemia (Endocrine disorders) | 2 (2)
Hyperkalemia (General disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (4)
Hypocalcemia (General disorders) | 1 (1)
Hypokalemia (General disorders) | 1 (1)
Hypomagnesemia (General disorders) | 1 (1)
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased liver function tests (Hepatobiliary disorders) | 1 (2)
Infection (Infections and infestations) | 1 (1)
Lethargy and confusion (General disorders) | 1 (1)
Neuropathic extremity pain (Nervous system disorders) | 1 (1)
Post transplant lymphoproliferative disorder (Surgical and medical procedures) | 1 (1)
Prograf toxicity (Surgical and medical procedures) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Vascular disorders) | 1 (1)
Rectal pain (General disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 2 (4)
Severe itching (General disorders) | 1 (1)
Severe pain (General disorders) | 1 (1)
Somnolence, depressed level of consciousness (General disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 7 (10)
Tremors (General disorders) | 1 (1)
Urinary disorder (Renal and urinary disorders) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (1)
Increased white blood cell count (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes